CLINICAL TRIAL: NCT01032759
Title: Memantine for Postoperative Analgesia
Brief Title: Memantine and Postoperative Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00019279
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Active Comparator)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — 20 mg, BID
  Arms: Memantine
Drug: Placebo — BID
  Arms: Placebo

SUMMARY:
Memantine is associated with improvement in pain relief after surgery.

DETAILED DESCRIPTION:
This prospective, randomized, controlled trial will investigate whether perioperative memantine has a postoperative analgesic effect following radical retropubic prostatectomy (RRP). 100-110 patients scheduled to undergo RRP at Duke will be assessed preoperatively for allodynia using Von Frey filaments, then stratified into two groups based on the presence or absence of allodynia. Patients in each group will then be randomized to receive either memantine 20 mg or placebo 30-60 minutes preoperatively, followed on postoperative day 1 with either memantine 10 mg in the morning and 10 mg in the evening for memantine patients, or placebo at the same intervals for placebo patients. Data such as morphine consumption, patient satisfaction and pain scores, opioid-related side effects, and the area of hyperalgesia around the surgical incision will be recorded for the initial 48 hours postoperatively, and patient satisfaction with their postoperative analgesia will be assessed after 1 week. At 1, 3, and 6 months postoperatively, patients will be asked about the presence and intensity of any persistent pain related to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18 to 75 years old

Exclusion Criteria:

* Chronic pain conditions or taking regular analgesics
* Taking psychotropic medications
* Parkinson's disease
* Narrow-angle glaucoma
* Known gastroduodenal ulcer
* History of seizure disorder
* Renal insufficiency, as defined by serum creatinine greater than 2 mg/dL
* Liver disease, including liver failure, cirrhosis, or acute hepatitis
* Significant coronary vascular disease or cardiac conduction system disease, as noted by ECG or history of cardiac symptoms, or cardiac ejection fraction less than 30%
* American Society of Anesthesiologists (ASA) score of 4 or higher
* Allergy to ketorolac or memantine

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 participants signed consent, 63 participants were randomized
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 32 | 31
Completed 24 Hour Assessment | 32 | 30
Completed 48 Hour Assessment | 31 | 28
Completed | 31 | 28
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (7) | 59 (7) | 59 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 31 | 63
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63

OUTCOME MEASURES:

1. Secondary Outcome: Pain Scores
Description: Pain score (0=no pain, 10= worst possible pain)
Time Frame: 48 hours
Population: Participants who completed the 48 hour assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 31 | 28
units on a scale | 2.64 (0.46) | 1.71 (0.40)

2. Primary Outcome: 24 hr Opioid Consumption
Time Frame: 24 hr
Population: Participants who completed the 24 hour assessment.
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 32 | 30
mg morphine equivalents | 21.5 (3.9) | 18.6 (4.0)

3. Secondary Outcome: Opioid Related Side Effects
Description: Number of participants with postoperative nausea and vomiting.
Time Frame: 0-24 h
Measure: Number; unit: participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 32 | 30
participants | 19 | 19

4. Secondary Outcome: Opioid Related Side Effects: Pruritus
Description: Number of participants who experienced pruritus.
Time Frame: 0-24 h
Measure: Number; unit: participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 32 | 30
participants | 7 | 9

5. Secondary Outcome: Hyperalgesia
Description: Stimulation with a Von Frey hair filament at 396 mN of force will be started from outside the hyperalgesic area, where no pain sensation is experienced toward the incision until the patient reports a distinct change in perception. The first point where a "painful," "sore," or "sharper" feeling occurs will be marked, and the distance to the incision measured. The surface area will be measured in cm2 around the surgical incision.
Time Frame: Within 48 h
Population: Number of participants who had this outcome measured and documented
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 20 | 19
cm2 | 56 (37) | 54 (36)

6. Secondary Outcome: Patient Satisfaction
Description: Number of participants who reported "very satisfied" or "somewhat satisfied"
Time Frame: 48 hours
Population: Number of participants who had this outcome reported and documented.
Measure: Number; unit: participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 32 | 30
participants | 30 | 25

7. Secondary Outcome: Chronic Post-surgical Pain
Time Frame: 1 month, 3 month, 6 month
Population: Data was not collected and therefore not analyzed.
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/31
Other Adverse Events (participants affected / at risk) | 0/32 | 1/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=32) | Placebo (N=31)
TIA (Nervous system disorders) | 1 (1) | 0 (0) — Transient ischemic attack
Pulmonary embolism (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=32) | Placebo (N=31)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes